CLINICAL TRIAL: NCT03879967
Title: Lateral Ridge Augmentation Using Allograft Blocks and Guided Bone Regeneration for Implant Sites
Brief Title: Lateral Ridge Augmentation Using Allograft Blocks and GBR for Implant Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allo_3_OCS_zmkUnibe
Record Dates: First submitted 2019-03-08; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Alveolar Ridge Augmentation
Keywords: Allograft block; guided bone regeneration; implants

STUDY DESIGN:
Intervention Model Description: A group of thirteen patients were selected for lateral ridge augmentation using cortico-cancellous allogenic block with guided bone regeneration. After the first surgery a healing phase was given and then a second surgery for implant placement in these augmented sites was carried out. Post healing, the implants were prosthetically restored and followed up upto three years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allograft block graft (Experimental): For lateral alveolar ridge augmentation, all patients will be treated with allograft block with guided bone regeneration. After a minimal healing phase of six months, implants would be placed in the augmented site. After a healing phase of about 4months, the implants would be loaded and then followed until the control appointment approximately 3 years later.
  Interventions: Device: Allograft block graft

INTERVENTIONS:
Device: Allograft block graft — The graft used is a mineralized, cortico-cancellous, delipidized, lyophilized allogenic block.

SUMMARY:
Clinicians are increasingly faced with the challenge of reconstructing the alveolar ridge as more patients desire fixed implant-supported restorations. Reconstruction of large horizontal alveolar defects still remains a challenge in implantology. Although autogenous blocks from intraoral sites are proven effective for such defects, donor site morbidity and limited graft availability are major limitations. Allogenic bone blocks have been proposed to overcome these limitations, however, the outcomes reported in the literature are inconclusive. In this case series, the efficacy of allogenic blocks for lateral augmentation of atrophic ridges was evaluated, over a three-year period.

In nineteen edentulous sites from ten patients, cortico-cancellous allogenic blocks (PHOENIX, TBF, France) were shaped to the defect and screw-fixated. A double-layer of autogenous chips and demineralized bovine bone (Bio-Oss, Geistlich Pharma AG, Switzerland) was used to fill the voids. The augmented site was covered by non-cross-linked collagen membrane (Bio-Gide, Geistlich Pharma AG, Switzerland). After a healing period of 9 months, implants were placed and CBCT analysis was performed post-implantation. Following a period of 34 months of function (range 22 to 44 months), patients were clinically and radiographically re-examined.

DETAILED DESCRIPTION:
The present study design is a mono-center three-year follow-up case series study to examined the safety and effectiveness of allograft bone blocks combined with guided bone regeneration (GBR). The study was in accordance to the principles of the Declaration of Helsinki and was approved by the standing ethical committee of the state of Bern, Switzerland.

The preoperative analysis included a complete medical history, clinical examination of the dentition and a thorough analysis of the implant recipient using 3D cone beam computed tomography (3D Accuitomo 170, Morita, Kyoto, Japan).

Surgical Procedure:

The surgical procedures were done in two stages. In the first stage surgery, a full-thickness mucoperiosteal flap was raised on both the facial and palatal aspects. Ridge augmentation was done using a mineralized, cortico-cancellous, delipidized, lyophilized allogenic block (ALB ; PHOENIX allograft, TBF Mions, France). Following hydration of the ALB, the cortico-cancellous part of the block was shaped to fit the recipient site and fixated by two fixation screws (Medartis, Modus, Medartis Holding AG, Basel, Switzerland). Voids around the ALB were filled with autogenous bone chips (AGB) harvested locally from the recipient site. The augmented site was covered by a first layer of deproteinized bovine bone mineral mixed (DBBM; Bio- Oss, Geistlich Pharma, Wolhusen, Switzerland and a non-crosslinked collagen membrane (BG; Bio- Gide, Geistlich AG, Wolhusen, Switzerland) as described previously (Chappuis et al DOI 10.1111/cid.12438). A periosteal-releasing incision was used to provide tension-free flap closure. The wound margins were approximated using non-resorbable poly- amide suture (Seralon, Serag-Wiessner GmbH, Naila, Germany) to obtain primary wound closure. All patients were prescribed an antibiotic regimen with 2g of amoxicillin with clavulanic acid 1 hour preoperatively to be continued as 1g twice daily for 3 days post-surgery. Patients were also prescribed analgesics and chlorhexidine digluconate (0.2%) for chemical plaque control. In patients with post-surgical complications the antibiotic regimen was prolonged. Sutures were removed around 14 days postoperatively. Removable provisionals were adapted, but patients were instructed to not to wear them unless unavoidable during the initial healing phase.

The second stage surgery was performed after a minimal healing period of six months (range 6 to 13months for me this would belong to the results). A paracrestal incision was given to elevate a full thickness mucoperiosteal. The fixation screws from the previous surgery were removed and the implant bed was prepared based on the specific requirements of the site. All implants placed had chemically modified, sandblasted, and acid-etched surface and had either, a tissue level implant (TL) or a bone level implant (BL) design (SLActive, Straumann AG, Basel, Switzerland). Simultaneous re-grafting was performed as required using autogenous bone chips, DBBM and a non-cross linked collagen membrane. A tension-free wound closure was obtained by non-resorbable sutures. The antibiotic and analgesic regimen and post-surgical care as the same as in the first-stage surgery. Sutures were removed after 14 days. Patients were instructed to wear the provisional with caution. After the healing period of 4-6 months the healing abutments were placed for the future prosthetics. The implants were restored with either single-unit crowns (SC), crowns with extensions (SC-E), bridges (B), bridges with extensions (B-E) or ball abutments (BA). All restorations were screw-retained. Patient were given oral hygiene instructions and directed to enroll onto a supportive periodontal therapy to monitor oral health.

Clinical and radiographic follow-up examination after 3 years:

Clinical parameters - Updates on medical conditions, smoking, oral hygiene and enrollment in a maintenance care program were collected from the patients. Clinical examinations were taken by the same examiner (VC) throughout the three-year follow-up period. The clinical parameters were assessed as previously described (Chappuis et al DOI 10.1111/cid.12438): peri-implant suppuration, modified plaque index (mPLI), modified sulcus bleeding index (mBLI), probing depth, DIM (distance from the implant shoulder to the mucosal margin), width of the KM, mobility and full mouth plaque scores.

Radiographic analysis using 2D radiographs and 3D CBCT - The peri-implant bone loss was measured on periapical 2D radiographs analysing the proximal DIB values as the vertical distance from the implant shoulder to the first bone-to-implant contact as described earlier (DIB; mm) (Weber HP et al 1992). The mean DIB value per implant considered was the average of the mesial and distal values.

The horizontal bone gain of the atrophic sites was assessed by with the smallest field of view (3D Accuitomo 170, Morita, Kyoto, Japan). The image analysis was performed by a high-resolution screen, using a specialised software (i-Dixel, Morita, Kyoto, Japan). The 3D analysis included a preoperative analysis of the proposed implant site. A standard reference point, 4mm crestal to the shoulder of the future implant was used for all measurements (Chappuis 2017). CBCT measurements were repeated prior to implant placement, using the same reference point and repeated again at the 2-3year follow-up appointment. The radiographic measurements were done by one examiner (OE).

Assessment of biological, technical complications and patient reported outcome measures (PROMS) - All events of complications, intra-operative and post-operative at each surgical phase (graft surgery and implant surgery), prior to prosthetic treatment and post prosthetic rehabilitation both operator-assessed and self-reported were recorded.

Patient reported outcome measures were assessed by the Oral Health Impact Profile (OHIP) scores and patient satisfaction scores based on a visual analog scale (VAS) were recorded for each patient after the entire treatment was completed and the patients received the prosthetic replacements.

Statistical Analysis:

All data sets were first analysed descriptively and were expressed as mean values with standard deviation. A repeated measures design was chosen and a linear mixed model was fitted for each single factor to assess its impact on the final outcome and co-relations were evaluated. Throughout, p-values less than 0.05 were considered as statistically significant. p-values were not corrected for multiple testing due to the explorative nature of this study. The statistical analysis was performed with the software package R (Version 3.5.1, R Foundation for Statistical Computing, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

1. Atrophy of the alveolar ridge in the horizontal plane (<4 mm in posterior sites and <5 mm in anterior sites), or a crest width 5 mm in esthetic sites.
2. Patients who agree to sign an informed consent.

Exclusion Criteria:

1. Patients who had adequate horizontal ridge thickness and did not require ridge augmentation
2. Patients with deficient vertical height of the ridge requiring vertical augmentation
3. Patients who were not ready for implant supported prosthesis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Change in ridge thickness with use of the allograft block | The measurements were done at approximately 9 months after ridge augmentation surgery and prior to implant placement.
  The change in ridge thickness was measured in mm at a specific reference point 4mm apical to the shoulder of the implant. The measurements were done from a CBCT image in the coronal/sagittal plane.
Change in ridge thickness with use of the allograft block after implant placement | The measurements were done at the follow-up appointment approximately 3years after implant placement.
  The change in ridge thickness was measured in mm at a specific reference point 4mm apical to the shoulder of the implant. The measurements were done from a CBCT image in the coronal/sagittal plane.

SECONDARY OUTCOMES:
Peri-implant suppuration | Recorded at the 3years follow-up time point
  Measured by palpation and probing
Modified plaque index by Mombelli | Recorded at the 3years follow-up time point
  Measured visually and with a periodontal probe. Assessed at four aspects around the implants mesial, distal, buccal and lingual.
  score 0, no detection of plaque; score 1, plaque only recognized by running a probe across the smooth marginal surface of the implant; score 2, plaque can be seen by the naked eye; and score 3, abundance of soft matter. The average of the four scores, gives the Modified plaque index for the implant
Modified sulcus bleeding index by Mombelli | Recorded at the 3years follow-up time point
  Measured visually and with a periodontal probe.Measured visually and with a periodontal probe. Assessed at four aspects around the implants mesial, distal, buccal and lingual.
  score 0: no bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant; score 1: isolated bleeding spot visible; score 2: blood forms a confluent red line on margin; score 3: heavy or profuse bleeding. The average of the four scores gives the Modified sulcus bleeding index for the implant
Probing depth | Recorded at the 3years follow-up time point
  Measured with a periodontal probe in mm. Normal probing depth is between 1-3mm.
Distance from the implant shoulder to the mucosal margin | Recorded at the 3years follow-up time point
  Measured in mm from a 2D radiograph on mesial and distal aspects of the implant
Width of the keratinized mucosa | Recorded at the 3years follow-up time point
  Measured with a probe in mm on the buccal surface
Mobility | Recorded at the 3years follow-up time point
  Measured by palpation and resonance frequency analysis. Resonance frequency value les than 60 shows low stability and over 70 shows high stability.
Full mouth plaque scores | Recorded at the 3years follow-up time point
  Full mouth plaque score expressed as a percentage
Number of participants with intraoperative complications at graft surgery | During graft surgery
  Presence or absence of intraoperative complications as assessed by operator. Score 1 : no complications score 2: bleeding The patient is allotted one of the two scores
Number of participants with intraoperative complications at implant surgery | During the implant placement surgery
  Presence or absence of intraoperative complications as assessed by operator. Score 1 : no complications score 2: bleeding The patient is allotted one of the two scores
Number of participants with post graft surgery complications | One day after to 6 months post graft surgery
  Presence or absence of post surgical complications as assessed by operator or reported by patient score 1: no complication score 2: hematoma score 3: post operative bleeding score 4: infection score 5: sequestrum The implant is allotted one of the above scores
Number of participants with post implant surgery complications | One day after to 6 months post implant surgery
  Presence or absence of post surgical complications as assessed by operator or reported by patient score 1: no complication score 2: hematoma score 3: post operative bleeding score 4: infection score 5: sequestrum The implant is allotted one of the above scores
Number of patients with technical complications | One day after to 3 months post prosthetic rehabilitation
  Presence of absence of technical complications with prosthesis as assessed by operator or reported by patient.
  score 1: no complication score 2: chipping score 3: framework fracture score 4:loosening score 5: abutment fracture score 6: new crown to be fabricated The implant is allotted one of the above scores
Visual Analog Scale | 3 years afer implant placement
  As assessed by the patient to rate the experience with the prosthesis on a scale of 1 to 100 with 1 being the lowest and 100 being the highest score
Oral Health Impact Profile 14 | 3 years after implant placement
  As assessed by the patient to rate the overall treatment. The patient has to answer 14 questions related to the treatment and each question is scored from a score of 0 to 4.
  score 0: never, score l: hardly ever score 2: occasionally score 3: fairly often, score 4: very often The scores for all questions are added to obtain a score for the patient

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Buser Prof, DDS,DMD, Study Chair — Department of Oral Surgery and Stomatology, ZMK, University of Bern; Vivianne Chappuis Prof, PD, DMD, Study Director — Department of Oral Surgery and Stomatology, ZMK, University of Bern; Odette Engel, Dr med dent, Principal Investigator — Department of Oral Surgery and Stomatology, ZMK, University of Bern; Supriya Ebenezer, BDS, MDS, Principal Investigator — Department of Oral Surgery and Stomatology, ZMK, University of Bern
Locations (1):
- Department of Oral Surgery and Stomatology, ZMK, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chappuis V, Cavusoglu Y, Buser D, von Arx T. Lateral Ridge Augmentation Using Autogenous Block Grafts and Guided Bone Regeneration: A 10-Year Prospective Case Series Study. Clin Implant Dent Relat Res. 2017 Feb;19(1):85-96. doi: 10.1111/cid.12438. Epub 2016 Jul 31. PMID 27476677

DOCUMENTS (1):
  • Study Protocol (2018-12-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT03879967/Prot_000.pdf